CLINICAL TRIAL: NCT02435706
Title: Esthetic Outcomes of Single Immediate Implant Placement With Immediate Restoration Performed With Two Surgical Techniques
Brief Title: Esthetic Outcomes of Single Immediate Implant Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Elena Sanz Miralles, Assistant Professor of Dental Medicine (Periodontics), Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAI1840
Record Dates: First submitted 2015-04-15; First posted 2015-05-06 (Estimated); Results first posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-04

CONDITIONS: Gingival Recession; Bone Loss, Alveolar
Keywords: Dental implants; surgical flap; esthetics; alveolar process
MeSH Terms: conditions — Gingival Recession; Alveolar Bone Loss | interventions — Mutagenesis, Insertional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flapless immediate implant placement group (Experimental): Flapless placement of immediate implant and temporary crown
  Interventions: Procedure: Flapless immediate implant placement; Device: Implant and temporary crown
- Flap assisted immediate implant placement group (Active Comparator): Flap elevation prior to placement of immediate implant and temporary crown
  Interventions: Procedure: Flap assisted immediate implant placement; Device: Implant and temporary crown

INTERVENTIONS:
Procedure: Flapless immediate implant placement — Experimental group: No elevation of flap prior to immediate implant placement
  Arms: Flapless immediate implant placement group
Procedure: Flap assisted immediate implant placement — Control group: Flap will be elevated prior to immediate implant placement
  Arms: Flap assisted immediate implant placement group
Device: Implant and temporary crown — Both groups receive this intervention

SUMMARY:
A randomized controlled trial of 12-month duration to compare gingival margin location, buccal horizontal ridge dimensions, and interproximal crestal bone levels following two surgical approaches for immediate placement of implants in the esthetic zone: one involving flap elevation and another using a flapless protocol.

DETAILED DESCRIPTION:
In the test group, the implant will be placed according to standard protocol at a position engaging the palatal wall without elevation of a mucoperiosteal flap.

In the control group, intrasulcular incisions will be carried out from one tooth distal to one tooth mesial to the extraction site and full thickness flaps will be elevated with periosteal elevator, including the papillae. The implant will be placed according to standard protocol at a position engaging the palatal wall, and the flaps will be sutured using a combination of interrupted and mattress sutures.

In both groups, temporary restorations will be delivered immediately after implant placement provided that the implant shows primary stability and has engaged in the bone with an insertion torque of 25Ncm or more. In case of a lower insertion torque, the protocol will be abandoned, a cover screw will be placed, and a two stage implant protocol will be followed. All patients will be advised to receive a permanent restoration 6 months after surgery, if the implant is deemed to be successful.

ELIGIBILITY:
Inclusion Criteria:

* Single non-restorable tooth in the anterior maxilla
* Intact buccal plate or <5mm fenestration

Exclusion Criteria:

* Pregnancy
* Current smokers >10 cigarettes/day
* Parafunctional habits
* Malocclusion or intent of orthodontic therapy in the future
* Severe periodontal disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-12; Primary Completion 2016-08-09 (Actual); Study Completion 2016-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Sanz Miralles, DDS, MS, PhD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: Yes
De-identified data were shared with The University of Texas Science Center at Houston (Dr. Chun-Teh Lee, formerly at Columbia University) in order to pursue further analysis of the data.
Time Frame: April 2018. Data to be shared until the completion of the analysis of the data and publication of the results.
Access Criteria: De-identified data corresponding to clinical and radiographic measurements were shared. Data were shared with Dr. Chun-teh Lee, a former investigator of the study who is currently working at The University of Texas Science Center at Houston.

REFERENCES:
- [Background] Stoupel J, Lee CT, Glick J, Sanz-Miralles E, Chiuzan C, Papapanou PN. Immediate implant placement and provisionalization in the aesthetic zone using a flapless or a flap-involving approach: a randomized controlled trial. J Clin Periodontol. 2016 Dec;43(12):1171-1179. doi: 10.1111/jcpe.12610. Epub 2016 Oct 17. PMID 27501953
- [Background] Lee CT, Chiu TS, Chuang SK, Tarnow D, Stoupel J. Alterations of the bone dimension following immediate implant placement into extraction socket: systematic review and meta-analysis. J Clin Periodontol. 2014 Sep;41(9):914-26. doi: 10.1111/jcpe.12276. Epub 2014 Jul 23. PMID 24894299

RESULTS

PARTICIPANT FLOW:
Groups:
- Flapless Group: Flapless immediate implant placement: Flapless placement of immediate implant and temporary crown
  Flapless immediate implant placement: No elevation of flap prior to immediate implant placement
  Implant and temporary crown: Standard intervention/procedure (non-experimental)
  Please see attached publication
- Flap Group: Flap assisted immediate implant placement: Flap elevation prior to placement of immediate implant and temporary crown
  Flap assisted immediate implant placement: Flap will be elevated prior to immediate implant placement
  Implant and temporary crown: Standard intervention/procedure (non-experimental)
Period: Overall Study
Arm/Group | Flapless Group | Flap Group
Started | 18 | 21
Completed | 16 | 20
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Flapless Group: Flapless immediate implant placement: Flapless placement of immediate implant and temporary crown
  Flapless immediate implant placement: No elevation of flap prior to immediate implant placement
  Implant and temporary crown: Standard intervention/procedure (non-experimental)
- Total: Total of all reporting groups
Arm/Group | Flapless Group | Flap Group | Total
Number analyzed (Participants) | 18 | 21 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 17 | 30
  >=65 years | 5 | 4 | 9
Age, Continuous [Median (Full Range); unit: years] | 54 [20 to 85] | 46 [22 to 73] | 48 [20 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 8 | 6 | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 21 | 39

OUTCOME MEASURES:

1. Primary Outcome: Change in Gingival Margin Location on the Buccal, Mesial and Distal Compared With Pre-operative Baseline and Post-operative Baseline
Time Frame: Change from Pre-operative Baseline in Gingival Margin Location at 3, 6 and 12 months and change from post-operative baseline at 3 and 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Flapless Group | Flap Group
Number analyzed (Participants) | 18 | 21
mm
  From pre-operative to 3 months follow-up (Mesial) | .11 (0.32) | .43 (.37)
  From pre-operative to 3 months follow-up (Buccal) | .28 (.39) | .48 (.50)
  From pre-operative to 3 months follow-up (Distal) | .11 (.32) | .48 (.44)
  From pre-operative to 6 months follow-up (Mesial) | .11 (.32) | .40 (.48)
  From pre-operative to 6 months follow-up (Buccal) | .19 (.30) | .40 (.60)
  From pre-operative to 6 months follow-up (Distal) | .14 (.29) | .23 (.47)
  From pre-operative to 12 months follow-up (Mesial) | .09 (.27) | .22 (.43)
  From pre-operative to 12 months follow-up (Buccal) | .22 (.31) | .42 (.52)
  From pre-operative to 12 months follow-up (Distal) | .06 (.25) | .28 (.39)
  From post-operative to 3 months (Mesial) | -.25 (.46) | .10 (.48)
  From post-operative to 3 months (Buccal) | -.22 (.31) | .2 (.62)
  From post-operative to 3 months (Distal) | -.31 (.57) | 0 (.61)
  From post-operative to 6 months (Mesial) | -.50 (.54) | -.05 (.54)
  From post-operative to 6 months (Buccal) | -.25 (.39) | .13 (.60)
  From post-operative to 6 months (Distal) | -.25 (.73) | -.03 (.64)

2. Secondary Outcome: Change in Buccal Horizontal Ridge Dimensions
Description: Horizontal changes of the buccal ridge was calculated through the use of acrylic stents and digital overlays (3Shape D800, Biomet 3i, Palm Beach Gardens, FLS). The acrylic stents were obtained from the pre-surgical plaster casts and they were repositioned on the plaster casts obtained at 3, 6 and 12 months. Discrepancies between the acrylic stent and the plaster cast were measured with a probe. The digital cast overlays were used to analyze changes from pre-surgical to 3 and from 3 to 6 months). The plaster casts were scanned and changes were analyzed with the use of a software.
Time Frame: Change from Baseline in Buccal Horizontal Ridge Dimensions at 3, 6 and 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Flapless Group | Flap Group
Number analyzed (Participants) | 18 | 21
mm
  Casts(Digital Over delays) 0-3 months | .64 (.59) | .54 (.63)
  Casts(Digital Over delays) 3-6 months | .18 (.46) | .19 (.7)
  Casts (stents) 0-3 months | .58 (.60) | .80 (.83)
  Casts (stents) 0-6 months | .89 (.80) | .95 (.92)
  Casts (stents) 0-12 months | .91 (.84) | 1.11 (.92)

3. Secondary Outcome: Change in Interproximal Crestal Bone Levels
Time Frame: Change from Baseline in Interproximal Crestal Bone Levels at 6 and 12 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Flapless Group | Flap Group
Number analyzed (Participants) | 18 | 21
mm
  Bone level change at 6 months (mesial) | .31 (.47) | .37 (.91)
  Bone level change at 6 months (distal) | .45 (.81) | .82 (.87)
  Bone level change at 12 months (mesial) | .47 (.98) | .73 (1.18)
  Bone level change at 12 months (distal) | .59 (1.05) | 1.33 (1.23)

ADVERSE EVENTS:
Arm/Group | Flapless Group | Flap Group
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/21
Other Adverse Events (participants affected / at risk) | 0/18 | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Flapless Group (N=18) | Flap Group (N=21)
Early implant failure (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-28): https://cdn.clinicaltrials.gov/large-docs/06/NCT02435706/Prot_SAP_000.pdf